CLINICAL TRIAL: NCT02248389
Title: Evaluation of a Laparoscopic High Intensity Focused Ultrasound Probe for the Ablation of Small Renal Masses
Acronym: HIFU-KIDNEY
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: SonaCare Medical (Industry)
Responsible Party: Principal Investigator, Chandru Sundaram, Professor of Urology, Director of Minimally Invasive Surgery, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IUCRO-0474
Record Dates: First submitted 2014-09-19; First posted 2014-09-25 (Estimated); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Carcinoma, Renal Cell
Keywords: carcinoma, renal cell; ablation; laparoscopic surgery; high intensity focused ultrasound
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ablation arm (Experimental): Each person in study will receive ablation of their renal tumor followed by standard partial nephrectomy.
  Interventions: Device: Sonatherm 600i ablation system

INTERVENTIONS:
Device: Sonatherm 600i ablation system — HIFU ablation of tumor.

SUMMARY:
The Sonatherm device provides both advanced imaging (ultrasound guidance) and high intensity focused ultrasound to target and ablate tumors. It also does not require piercing the tumor with a needle as does cryotherapy (Cryo) and radiofrequency (RF) ablation. Cryo and RF also have high retreatment rates due the finding of untreated tumor on follow-up imaging. Thus, there is reason to hypothesize that Sonatherm with it's real-time ultrasound imaging feedback could replace RF and Cryo for the treatment of small renal masses where the invasiveness of full resection partial nephrectomy is contraindicated due to patient comorbidities.

DETAILED DESCRIPTION:
This study uses a treat and resect model where ablation is followed by a partial nephrectomy. This will allow for the ablation to be evaluated for necrosis and targeting accuracy. It will also ensure cancer safety prior validation of the HIFU device. The applied heat of HIFU ablation could improve hemostasis and blood loss.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age.
2. Must provide written informed consent
3. Must have presence of an enhancing solid renal mass ≤ 3.0 cm on CT or MRI
4. Must be scheduled for laparoscopic robot assisted partial nephrectomy of renal mass.
5. Must have an expected survival status of at least 3 months.
6. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1.
7. Previous chemotherapy, and/or biological therapy for cancer are permitted. The subject should have recovered from the effects of these or of any prior surgery.
8. Women of child bearing potential must have negative pregnancy test (urine or serum) prior to study enrollment. Females must agree to adequate birth control if conception is possible during the study.
9. All toxicities from prior therapy must be recovered to a grade 1 or better according to the Clavien-Dindo Classification system.
10. If previous biopsy of mass has been done, pathology must be consistent with renal cell carcinoma (RCC).

Exclusion Criteria

1. < 90% solid component of the tumor on screening cross-sectional imaging (CT/MRI)
2. Prior ablative or surgical treatment of the lesion
3. Masses located close to the hilar vessels or at locations that cannot be accessed with the HIFU probe
4. The patient has only one kidney
5. Multiple or bilateral renal masses
6. Failure to meet the following laboratory levels on preoperative screening:

   1. Platelet count ≥ 100,000 mm3
   2. Hemoglobin ≥ 10 g/dl.
   3. Prothrombin Time (PT) ≤ 1.5 times upper limit of laboratory normal (ULN).
   4. Activated partial thromboplastin time (aPTT) ≤ 1.5 times ULN.
   5. Serum creatinine < 2.5 times ULN.
7. Hepatic toxicity grade 2 (using CTCAE version 4 standard definitions)
8. Inability to hold anticoagulation for surgery due to high risk of a cerebral vascular event, myocardial event, or like risk (ASA may be continued)
9. Abdominal obesity that would, in the assessment of the PI, make the HIFU ablation difficult
10. Participation in another investigational trial concurrently or within 30 days prior to enrollment
11. Subjects with a diagnosis of metastatic disease who are currently receiving treatment or who are not in remission
12. Significant acute or chronic medical, neurologic, or psychiatric illness in the subject that, in the judgment of the Principal Investigator, could compromise subject safety, limit the subject's ability to complete the study, and/or compromise the objectives of the study

    -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-09-04 (Actual); Primary Completion 2015-06-08 (Actual); Study Completion 2015-06-08 (Actual)

PRIMARY OUTCOMES:
Operative and postoperative complications | 4-months
  Observing complications as defined by the Clavien system (1-5).

SECONDARY OUTCOMES:
Necrosis | 1-week
  A microscopic analysis will be performed to assess necrosis within the ablation zone.
Tumor targeting | 1-week
  The ablation border beyond the tumor will be measured on pathologic analysis with success being defined as 1-10mm.
Surgeon rated ease of use | 1-week
  A questionnaire assessing the ease of use of the Sonatherm instrument will be given to the surgeon after each case.

CONTACTS AND LOCATIONS:
Locations (1):
- IU Health University Hospital, Indianapolis, Indiana, United States